CLINICAL TRIAL: NCT06398535
Title: Ultrasound Versus Magnetic Reseonance Imaging(MRI) in the Assessment of Anterior Knee Pain
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Asmaa Mostafa Abdelrady, Resident- Radiology department-sohag hospital university, Sohag University
Other Study IDs: soh-med-24-4-01MS
Record Dates: First submitted 2024-05-01; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Anterior Knee Pain
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: magenetic resonance and ultrasound — examination of patient using magentic resonace coil for imaging of knee and comapring the results obtaines by ultrasound examination using the ulatrsound tarsnsducer .

SUMMARY:
Anterior knee pain , often known as patellofemoral pain syndrome (PFPS), is a prevalent orthopedic ailment. It usually happens while you're bending your knees. It can affect people of all ages, although it is most common among teenagers, young adults, and athletes .

The actual etiology of anterior knee pain might be complicated, encompassing a variety of conditions; it causes disability, discomfort and a negative impact on the quality of life

. A number of diagnostic techniques, including plain radiography, computed tomography, MRI, arthroscopy and ultrasound are used to identify the pathologies causing anterior knee pain. Arthroscopy, though accurate, is invasive and can cause complications. Palin radiographs and computed tomography expose patients to radiations

ELIGIBILITY:
Inclusion Criteria:

* Adults who presented by knee pain , limitation of movement at knee.

Exclusion Criteria:

* Knee trauma, non-cooperative patients and those who refuse to participate, contraindications to magnetic resonance imaging, such as patients with cardiac pacemakers, metallic plates, and claustrophobia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Adults who presented by knee pain , limitation of movement at knee.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2024-12-10 (Estimated); Study Completion 2024-12-10 (Estimated)

PRIMARY OUTCOMES:
sensitivity | 6 months
  degress of sensitivity of ultrsound compaired to magentic resonance

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Crossley KM, Callaghan MJ, van Linschoten R. Patellofemoral pain. BMJ. 2015 Nov 4;351:h3939. doi: 10.1136/bmj.h3939. No abstract available. PMID 26537829
- [Background] Samim M, Smitaman E, Lawrence D, Moukaddam H. MRI of anterior knee pain. Skeletal Radiol. 2014 Jul;43(7):875-93. doi: 10.1007/s00256-014-1816-7. Epub 2014 Jan 29. PMID 24473994
- [Background] Sanchis-Alfonso V, Dye SF. How to Deal With Anterior Knee Pain in the Active Young Patient. Sports Health. 2017 Jul/Aug;9(4):346-351. doi: 10.1177/1941738116681269. Epub 2016 Nov 1. PMID 27920260
- [Background] Alves TI, Girish G, Kalume Brigido M, Jacobson JA. US of the Knee: Scanning Techniques, Pitfalls, and Pathologic Conditions. Radiographics. 2016 Oct;36(6):1759-1775. doi: 10.1148/rg.2016160019. PMID 27726755